CLINICAL TRIAL: NCT01331720
Title: Assessment of the Effectiveness and Tolerability of Ovarian Hyperstimulation Protocols Which Are the Most Common in Clinical Practice Using High Purified Gonadotrophins (u-FSH-HP y u-hMG-HP) in IVF/ICSI
Brief Title: Assessment of the Effectiveness and Tolerability of Ovarian Hyperstimulation
Acronym: DESCARTES
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring SAU (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Other Study IDs: FER-MEN-2006-03
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: STERILITY
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- FSH:LH 1:1 - Treatment Group A: Patients with a condition
  LH (luteinizing hormone)
  Interventions: Drug: hMG-HP
- FSH:LH 3:2 - Treatment Group B: Patients with a condition
  Interventions: Drug: hMG-HP
- FSH:LH 3:1 - Treatment Group C: Patients with a condition
  Interventions: Drug: hMG-HP
- FSH:LH 3:0 - Treatment Group D: Patients with a condition
  Interventions: Drug: hMG-HP
- Initially FSH:LH 3:0 and on S6 FSH:LH 1:1 - Treatment Group E: Patients with a condition
  Interventions: Drug: hMG-HP

INTERVENTIONS:
Drug: hMG-HP

SUMMARY:
The aim of the study is to assess the effectiveness of 5 mixed protocols of ovarian hyperstimulation with urinary gonadotrophins to achieve clinical pregnancy in females undergoing assisted reproductive techniques (IVF/ICSI) (in-vitro fertilisation/intracytoplasmic sperm injection).

Study hypothesis: mixed protocols with urinary FSH (follicle-stimulating hormone) and urinary hMG (human menopausal gonadotropin)should be more effective than monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30
* Prolactin within the laboratory normal range
* Couples affected by sterility able to treat by IVF/ICSI (in-vitro fertilisation/intracytoplasmic sperm injection)
* Patients undergoing Menopur® and/or Bravelle® treatment
* Normal thyroid function
* Women not receiving clomifen citrate or gonadotrophins within one month prior study start
* Couples willing to participate in the study that have signed the informed consent form

Exclusion Criteria:

* Failure in 3 previous cycles of assisted reproduction IVF/ICSI (in-vitro fertilisation/intracytoplasmic sperm injection)
* Policystic ovarian syndrome
* Seminal samples not apt for IVF-ICSI (according to the criteria of each center)
* Evidence of significant bacterial infection in the seminogram of the couple in the preceding 6 months
* Antecedents of severe ovarian hyperstimulation syndrome (OHSS)
* Important systemic disease
* Pregnancy or contraindication to pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females affected by sterility able to undergo IVF/ICSI
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 0-30 days

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 0-16 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (14):
- Spain (14):
  - Investigational site, Albacete, Albacete
  - Investigational site, Alicante, Alicante
  - Investigational site, Elche, Alicante
  - Investigational site, Badajoz, Badajoz
  - Investigational site, Castellon, Castellón
  - Investigational site, Santiago de Compostela, La Coruña
  - Investigational site, Mallorca, Mallorca
  - Investigational site, Murcia, Murcia
  - Investigational site, Málaga, Málaga
  - Investigational site, Navarra, Pamplona
  - Investigational site, Gijón, Principality of Asturias
  - Investigational site Sta. Cruz, Santa Cruz de Tenerife, Tenerife
  - Investigational site, Valencia, Valencia
  - Investigational site, Zaragoza, Zaragoza